CLINICAL TRIAL: NCT03800303
Title: Healthy Youth & Families: An Integrated Approach to Treating Mood Disorders
Brief Title: Integrated Treatment for Youth With Mood Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jarrod M. Leffler, Ph.D., L.P., Assistant Professor, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-010831
Record Dates: First submitted 2018-03-15; First posted 2019-01-11 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Mood Disorders in Children and Adolescents
Keywords: depression; bipolar; caregivers; children; adolescents; treatment; parents
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- two-week family-based treatment (Experimental): Active treatment includes a two-week family-based partial hospitalization treatment utilizing and integrated therapeutic design.
  Interventions: Behavioral: Family-based treatment

INTERVENTIONS:
Behavioral: Family-based treatment — 2-week family-based treatment

SUMMARY:
In an effort to understand the effects of evidence-based interventions on children and adolescents, the aims of this study are to:

1. evaluate the feasibility of utilizing wearable devices to track health information (i.e., sleep, physical activity);
2. evaluate the effectiveness of evidence-based intervention components on mood and interpersonal functioning, family engagement, and sleep and physical activity level outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents between the ages of 10 and 18 years;
* Diagnosed with a primary depressive or bipolar disorder;
* Admitted to the Child and Adolescent Integrated Mood Program (CAIMP) at Mayo Clinic.

Exclusion Criteria:

* Individual's not eligible for admission to the Child and Adolescent Integrated Mood Program (CAIMP)at Mayo Clinic.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Conner's Comprehensive Behavior Rating Scales | 12 months
  Likert scale items measuring symptom presentation

CONTACTS AND LOCATIONS:
Overall Officials: Jarrod M Leffler, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials